CLINICAL TRIAL: NCT00066170
Title: Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Parallel-Group, Multi-Center Trial Comparing the Effects of Orally Administered Xyrem (Sodium Oxybate) and Modafinil With Placebo in Treatment of Daytime Sleepiness in Narcolepsy
Brief Title: Trial Comparing Effects of Xyrem Taken Orally and Modafinil With Placebo in Treating Daytime Sleepiness in Narcolepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Senior Director Clinical Development, Jazz Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMC-SXB-22
Record Dates: First submitted 2003-08-04; First posted 2003-08-06 (Estimated); Results first posted 2011-11-30 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Narcolepsy
Keywords: Narcolepsy; Daytime Sleepiness; Daytime sleepiness in narcolepsy
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence | interventions — Sodium Oxybate; Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1. (Experimental): Xyrem + Modafinil Placebo
  Interventions: Drug: Xyrem; Drug: Modafinil (Placebo)
- Group 2: (Placebo Comparator): Xyrem Placebo + Modafinil Placebo
  Interventions: Drug: Xyrem Placebo; Drug: Modafinil (Placebo)
- Group 3 (Active Comparator): Xyrem Placebo + Modafinil at established dose
  Interventions: Drug: Xyrem Placebo; Drug: Modafinil at established dose
- Group 4: (Experimental): Xyrem + Modafinil at established dose
  Interventions: Drug: Xyrem; Drug: Modafinil at established dose

INTERVENTIONS:
Drug: Xyrem — Xyrem oral solution at 6 g/day for 4 weeks and 9 g/day for another 4 weeks.
  Other Names: Sodium Oxybate
  Arms: Group 1.; Group 4:
Drug: Xyrem Placebo — Xyrem Placebo oral solution 12 ml per day for 4 weeks and 18 ml per day for another 4 weeks.
  Other Names: Sodium Oxybate Placebo
  Arms: Group 2:; Group 3
Drug: Modafinil at established dose — Modafinil oral capsules at 200 to 600 mg per day for 8 weeks.
  Other Names: Provigil
  Arms: Group 3; Group 4:
Drug: Modafinil (Placebo) — Modafinil Placebo oral capsules 1 to 3 capsules per day for 8 weeks.
  Other Names: Provigil Placebo
  Arms: Group 1.; Group 2:

SUMMARY:
This study will be conducted as a randomized, double blind, double-dummy, placebo-controlled, parallel-group trial in patients diagnosed with narcolepsy. Volunteers for this trial will be required to make 5 visits over up to 14 weeks to a participating expert physician practitioner for various sleep and narcolepsy evaluations and diaries will also be collected. Participants will take assigned medications during the course of the trial. Subjects will have a 25% probability of receiving placebo for both drugs (modafinil and Xyrem). All subject volunteers must meet criteria for narcolepsy and have evidence of daytime sleepiness. Patients will not incur any personal medical expenses due to participation in this trial. The sponsor is covering all visit costs not covered by insurance and there are some funds for patient expenses such as travel.

ELIGIBILITY:
INCLUSION CRITERIA

Patients will be included in the trial if they:

* Have signed and dated an informed consent prior to beginning protocol required procedures.
* Are willing and able to complete the entire trial as described in the protocol.
* Are 18 years of age or older.
* Fulfill the International Classification of Sleep Disorders criteria for the diagnosis of narcolepsy.
* Are taking stable doses of modafinil (200 to 600 mg/day) for the treatment of daytime sleepiness for a period of three months or greater and the modafinil dose has been stable for at least 1 month prior to entering this trial
* Females may be included who are surgically sterile, two years post-menopausal, or if of child-bearing potential, using a medically accepted method of birth control (e.g., barrier method with spermicide, oral contraceptive, or abstinence) and agree to continue use of this method for the duration of the trial.
* In the opinion of the investigator have adequate support for the duration of the trial to include transportation to and from the trial site. In addition, if in the investigator's assessment it is clinically indicated, the patient is willing to not operate a car or heavy machinery for the duration of the trial or for as long as the investigator deems clinically indicated.

EXCLUSION CRITERIA

Patients will be excluded from the trial if they:

* Have received gamma-hydroxybutyrate in the last 30 days.
* Have taken any investigational therapy within the 30-day period prior to the initial screening visit (Visit 1) for this trial.
* Have sleep apnea syndrome, defined as an Apnea Index > 10 per hour or an AHI (Apnea Hypopnea Index) greater than 15 per hour, or have any other cause of daytime sleepiness, and have any other disorder(s) that can be considered a primary cause of excessive daytime sleepiness (e.g., severe periodic leg movement syndrome as determined by the investigator, sleep apnea, sleep deprivation).
* Are taking hypnotics, tranquilizers, antihistamines (except for non-sedating antihistamines), benzodiazepines or clonidine at the start of the baseline period. Patients taking anticonvulsants are not eligible to participate event if they are willing to washout anticonvulsants for the trial.
* Are experiencing any major illness, including unstable cardiovascular, endocrine, neoplastic, gastrointestinal, hematologic, hepatic, immunologic, metabolic, neurological (other than narcolepsy/cataplexy), pulmonary, and/or renal disease which would place the patient at risk during the trial or compromise the objectives outlined in the protocol.
* Have psychiatric disorders, major affective or psychotic disorders, or other problems that, in the investigator's opinion, would preclude the patient's participation and completion of this trial or compromise reliable representation of subjective symptoms.
* Have a current or recent (within one year) history of a substance use disorder including alcohol abuse as defined by the DSM-IV.
* Have a serum creatinine greater than 2.0 mg/dL, abnormal liver function tests (SGOT [AST] or SGPT [ALT] more than twice the upper limit of normal), or elevated serum bilirubin (more than 1.5 times the upper limit of normal), or pre-trial ECG results demonstrating clinically significant arrhythmias, greater than a first degree AV block or a history of myocardial infarction within the last six months.
* Have an occupation that requires variable shift work or routine night shift.
* Have a clinically significant history of seizure disorder either past or present, a history of clinically significant head trauma (i.e., concussion resulting in clinically significant loss of consciousness) or past invasive intracranial surgery, and are taking anticonvulsant medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2003-04; Primary Completion 2004-07 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanping Zheng, MD, Study Director — Jazz Pharmaceuticals, Inc
Locations (40):
- United States (36):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - St. Jude Medical Center -- Sleep Disorders Institute, Fullerton, California
  - Pacific Sleep Medicine Services, Inc., Los Angeles, California
  - Neuro-Therapeutics, Inc., Pasadena, California
  - Pacific Sleep Medicine Services, Inc., San Diego, California
  - Stanford Sleep Disorders Clinic, Stanford, California
  - Clinical Research Group of St. Petersburg, Inc., St. Petersburg, Florida
  - Peoria Pulmonary Associates, Ltd, Peoria, Illinois
  - The Center for Sleep and Wake Disorders/Midwest Neurology, Danville, Indiana
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Community Research & Sleep Management Institute, Crestview Hills, Kentucky
  - Chest Medicine Associates DBA -- Sleep Medicine Specialists, Louisville, Kentucky
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - Sleep Disorders Center -- Union Hospital of Cecil County, Elkton, Maryland
  - Sleep Medicine Associates of Maryland, Towson, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University Sleep Center, St Louis, Missouri
  - New Jersey Neuroscience Institute at JFK Medical Center, Edison, New Jersey
  - Sleep Disorders Center of Rochester, Rochester, New York
  - Strong Sleep Disorders Center, Rochester, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - ALL-TRIALS Clinical Research, LLC -- Summit Sleep Disorder, Winston-Salem, North Carolina
  - Cincinnati Clinic & Sleep Management Institute, Cincinnati, Ohio
  - Community Research Management Associates,Inc., Cincinnati, Ohio
  - CSC Research -- Grove City Sleep Diagnostic Center, Grove City, Ohio
  - Lehigh Valley Hospital Sleep Disorders Center, Allentown, Pennsylvania
  - Capital Region Sleep Disorder Center, Carlisle, Pennsylvania
  - Center for Sleep Medicine, Lafayette Hill, Pennsylvania
  - Lowcountry Lung and Critical Care, PA, Charleston, South Carolina
  - SleepMed of South Carolina, Columbia, South Carolina
  - SDHRF Clinical Research Center, Sioux Falls, South Dakota
  - Sioux Valley Clinic -- Pulmonary, Sioux Falls, South Dakota
  - Sleep Disorders Center, Sioux Falls, South Dakota
  - Bhupesh Dihenia, MD, Lubbock, Texas
  - SLEEP WALKER -- Sleep Disorders Center & Neurodiagnostics--Lung Diagnostics, Ltd., San Antonio, Texas
  - Vermont Medical Sleep Disorders Center, Inc., Essex Junction, Vermont
- France (2):
  - Hopital Pitie Salpetriere -- Federation des Pathologies du sommeil, Paris, Cedex 13
  - Centre du sommeil -- Hopital Gui de Chauliac, Montpellier, Cedex 5
- Psychiatrische Universitatsklinik, Regensburg, Germany
- Neurologische Poliklinik -- Universitats Spital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] A randomized, double blind, placebo-controlled multicenter trial comparing the effects of three doses of orally administered sodium oxybate with placebo for the treatment of narcolepsy. Sleep. 2002 Feb 1;25(1):42-9. PMID 11833860
- [Background] Scrima L, Hartman PG, Johnson FH Jr, Thomas EE, Hiller FC. The effects of gamma-hydroxybutyrate on the sleep of narcolepsy patients: a double-blind study. Sleep. 1990 Dec;13(6):479-90. doi: 10.1093/sleep/13.6.479. PMID 2281247
- [Background] Lammers GJ, Arends J, Declerck AC, Ferrari MD, Schouwink G, Troost J. Gammahydroxybutyrate and narcolepsy: a double-blind placebo-controlled study. Sleep. 1993 Apr;16(3):216-20. doi: 10.1093/sleep/16.3.216. PMID 8506453
- [Background] A 12-month, open-label, multicenter extension trial of orally administered sodium oxybate for the treatment of narcolepsy. Sleep. 2003 Feb 1;26(1):31-5. PMID 12627729
- [Result] Black J, Houghton WC. Sodium oxybate improves excessive daytime sleepiness in narcolepsy. Sleep. 2006 Jul;29(7):939-46. doi: 10.1093/sleep/29.7.939. PMID 16895262
- [Result] Black J, Pardi D, Hornfeldt CS, Inhaber N. The nightly use of sodium oxybate is associated with a reduction in nocturnal sleep disruption: a double-blind, placebo-controlled study in patients with narcolepsy. J Clin Sleep Med. 2010 Dec 15;6(6):596-602. PMID 21206549
- [Derived] Husain AM, Bujanover S, Ryan R, Scheckner B, Black J, Profant J. Incidence and duration of common, early-onset adverse events occurring during 2 randomized, placebo-controlled, phase 3 studies of sodium oxybate in participants with narcolepsy. J Clin Sleep Med. 2020 Sep 15;16(9):1469-1474. doi: 10.5664/jcsm.8530. PMID 32356515
- [Derived] Dauvilliers Y, Roth T, Guinta D, Alvarez-Horine S, Dynin E, Black J. Effect of sodium oxybate, modafinil, and their combination on disrupted nighttime sleep in narcolepsy. Sleep Med. 2017 Dec;40:53-57. doi: 10.1016/j.sleep.2017.07.030. Epub 2017 Oct 7. PMID 29221779
- See also: Xyrem Informational website with the package insert — http://www.xyrem.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Xyrem Placebo + Modafinil Placebo: Xyrem Placebo volume equivalent to 6 grams per day for the first 4 weeks and 9 grams per day for the remaining 4 weeks + Modafinil Placebo equivalent to prior dosage.
- Xyrem + Modafinil Placebo: Xyrem 6 grams per day for the first 4 weeks and 9 grams per day for the remaining 4 weeks + Modafinil Placebo equivalent to prior dosage.
- Xyrem Placebo + Modafinil at Established Dose: Xyrem Placebo volume equivalent to 6 grams per day for the first 4 weeks and 9 grams per day for the remaining 4 weeks + Modafinil at participant's prior dosage.
- Xyrem + Modafinil at Established Dose: Xyrem 6 grams per day for the first 4 weeks and 9 grams per day for the remaining 4 weeks + Modafinil at participant's prior dosage.
Period: Overall Study
Arm/Group | Xyrem Placebo + Modafinil Placebo | Xyrem + Modafinil Placebo | Xyrem Placebo + Modafinil at Established Dose | Xyrem + Modafinil at Established Dose
Started | 56 | 55 | 63 | 57
Intent to Treat | 55 | 50 | 63 | 54
Completed | 49 | 45 | 59 | 48
Not Completed | 7 | 10 | 4 | 9
Not completed — Adverse Event | 2 | 4 | 1 | 7
Not completed — Serious Adverse Event | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Non-Compliance with Trial Medicine | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 3 | 0 | 0 | 0
Not completed — Other | 1 | 5 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Xyrem Placebo + Modafinil Placebo | Xyrem + Modafinil Placebo | Xyrem Placebo + Modafinil at Established Dose | Xyrem + Modafinil at Established Dose | Total
Number analyzed (Participants) | 55 | 50 | 63 | 54 | 222
Age Continuous [Mean (Standard Deviation); unit: years] | 41.0 (13.35) | 35.1 (12.86) | 38.9 (15.62) | 38.9 (15.87) | 38.6 (14.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 24 | 31 | 29 | 115
  Male | 24 | 26 | 32 | 25 | 107
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 43 | 47 | 57 | 48 | 195
  Black | 11 | 2 | 5 | 3 | 21
  Asian | 0 | 1 | 0 | 0 | 1
  Hispanic | 1 | 0 | 0 | 1 | 2
  Other | 0 | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Daytime Sleep Latency as Measured by the Maintenance of Wakefulness Test (MWT)
Description: The Maintenance of Wakefulness Test consisted of four 20 minute tests of the patient's ability to remain awake in soporific conditions. The Mean change from baseline to week 8 in the average MWT number of minutes until sleep onset was the primary endpoint.
Time Frame: Baseline to Week 8
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Xyrem Placebo + Modafinil Placebo | Xyrem + Modafinil Placebo | Xyrem Placebo + Modafinil at Established Dose | Xyrem + Modafinil at Established Dose
Number analyzed (Participants) | 56 | 55 | 63 | 57
Minutes | -2.72 (4.535) | 0.58 (5.675) | -0.53 (4.358) | 2.68 (5.071)
Statistical Analysis 1: Comparison: Xyrem Placebo + Modafinil Placebo vs Xyrem + Modafinil Placebo; Test type: Superiority or Other; p < 0.001, Dunnett's
Statistical Analysis 2: Comparison: Xyrem Placebo + Modafinil Placebo vs Xyrem + Modafinil at Established Dose; Test type: Superiority or Other; p < 0.001, Dunnett's

ADVERSE EVENTS:
Arm/Group | Xyrem Placebo + Modafinil Placebo | Xyrem + Modafinil Placebo | Xyrem Placebo + Modafinil at Established Dose | Xyrem + Modafinil at Established Dose
Serious Adverse Events (participants affected / at risk) | 2/56 | 0/55 | 1/63 | 1/57
Other Adverse Events (participants affected / at risk) | 39/56 | 33/55 | 34/63 | 45/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xyrem Placebo + Modafinil Placebo (N=56) | Xyrem + Modafinil Placebo (N=55) | Xyrem Placebo + Modafinil at Established Dose (N=63) | Xyrem + Modafinil at Established Dose (N=57)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Psychotic Disorder due to a General Condition (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Xyrem Placebo + Modafinil Placebo (N=56) | Xyrem + Modafinil Placebo (N=55) | Xyrem Placebo + Modafinil at Established Dose (N=63) | Xyrem + Modafinil at Established Dose (N=57)
Vision Blurred (Eye disorders) | 1 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 12 | 2 | 12
Vomiting (Gastrointestinal disorders) | 0 | 7 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 3
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 3
Asthenia (General disorders) | 2 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 4 | 5 | 3 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 0
Headache (Nervous system disorders) | 12 | 5 | 7 | 11
Dizziness (Nervous system disorders) | 3 | 4 | 2 | 12
Somnolence (Nervous system disorders) | 4 | 4 | 2 | 3
Tremor (Nervous system disorders) | 0 | 3 | 0 | 8
Paraesthesia (Nervous system disorders) | 0 | 4 | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 0 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 1 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Keratoconjunctivitis Sicca (Eye disorders) | 0 | 2 | 0 | 1
Eye Discharge (Eye disorders) | 1 | 0 | 0 | 0
Eye Redness (Eye disorders) | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0
Visual Disturbance (Eye disorders) | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Loose Stools (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Aptyalism (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral Mucosal Disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary Hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue Blistering (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue Dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 1
Influenza like Illness (General disorders) | 0 | 2 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 1 | 1
Feeling Drunk (General disorders) | 0 | 1 | 1 | 1
Chest Pain (General disorders) | 0 | 0 | 1 | 1
Oedema Peripheral (General disorders) | 2 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 0
Application Site Dermatitis (General disorders) | 0 | 1 | 0 | 0
Chest Discomfort (General disorders) | 0 | 1 | 0 | 0
Feeling Cold (General disorders) | 0 | 0 | 0 | 1
Feeling Hot (General disorders) | 0 | 1 | 0 | 0
Feeling Hot and Cold (General disorders) | 0 | 0 | 0 | 1
Gait Abnormal (General disorders) | 0 | 1 | 0 | 0
Lethargy (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 1 | 0
Thirst (General disorders) | 1 | 0 | 0 | 0
Ulcer (General disorders) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 1 | 1
Sinusitis (Infections and infestations) | 3 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 2
Herpes Simplex (Infections and infestations) | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1
Adenoiditis (Infections and infestations) | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Dental Caries (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Back Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tooth Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Weight Increased (Investigations) | 3 | 0 | 1 | 0
White Blood Cell Count Increased (Investigations) | 0 | 1 | 0 | 1
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 0
Blood Glucose Abnormal (Investigations) | 0 | 0 | 0 | 1
Blood Lactate Dehydrogenase Abnormal (Investigations) | 0 | 0 | 1 | 0
Blood Potassium Decreased (Investigations) | 0 | 0 | 1 | 0
Eosinophil Count Increased (Investigations) | 0 | 0 | 0 | 1
Heart Rate Increased (Investigations) | 0 | 0 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 0 | 1 | 0 | 0
Lymphocyte Count Abnormal (Investigations) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Food Craving (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Cataplexy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Balance Disorder (Nervous system disorders) | 0 | 2 | 1 | 1
Ataxia (Nervous system disorders) | 1 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 1
memory Impairment (Nervous system disorders) | 1 | 0 | 0 | 1
Muscle Contractions Involuntary (Nervous system disorders) | 0 | 0 | 1 | 1
Sinus Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Burning Sensation (Nervous system disorders) | 0 | 1 | 0 | 0
Disturbance in Attention (Nervous system disorders) | 0 | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Hypertonia (Nervous system disorders) | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 1
Speech Disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Spinal Column Stenosis (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Tension Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 1 | 1 | 1
Disorientation (Psychiatric disorders) | 1 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 1
Crying (Psychiatric disorders) | 0 | 1 | 1 | 1
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 2
Nervousness (Psychiatric disorders) | 0 | 1 | 0 | 2
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 1 | 2
Affect Lability (Psychiatric disorders) | 0 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 0
Abnormal Dreams (Psychiatric disorders) | 0 | 0 | 0 | 1
Affective Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Belligerence (Psychiatric disorders) | 0 | 0 | 1 | 0
Dissociation (Psychiatric disorders) | 0 | 0 | 1 | 0
Euphoric Mood (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0
Impulsive Behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0
Libido Increased (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic Disorder due to a General Medical Condition (Psychiatric disorders) | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0
Sleep Attacks (Psychiatric disorders) | 0 | 1 | 0 | 0
Enuresis (Renal and urinary disorders) | 0 | 2 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Pollakiura (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hyperventialtion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal Passage Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatits Contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Oily Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hot Flush (Vascular disorders) | 1 | 0 | 2 | 1
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral Coldness (Vascular disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other